CLINICAL TRIAL: NCT05692050
Title: Expanded Access to Epcoritamab
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Other Study IDs: C23-496
Record Dates: First submitted 2023-01-13; First posted 2023-01-20 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection
  Other Names: ABBV-GMAB-3013

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to epcoritamab prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

- The participant must not be eligible for an epcoritamab clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie